CLINICAL TRIAL: NCT02907606
Title: Urinary Circulating Tumor DNA Detection in Non-small Cell Lung Cancer: a Prospective Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: San Valley Biotechnology Incorporated (Unknown)
Responsible Party: Principal Investigator, Jun Wang, Chief of Thoracic Department, Peking University People's Hospital
Other Study IDs: PKUPH-XW1401
Record Dates: First submitted 2016-09-08; First posted 2016-09-20 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Carcinoma; Non-small-cell Lung Cancer; Lung Neoplasms
Keywords: Non-small-cell Lung Cancer; circulating tumor DNA; urine
MeSH Terms: conditions — Carcinoma; Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Fresh tumor tissue, peripheral blood samples and urinary samples will be collected from each patient.
  Time:Preoperative, intraoperative, 3 days and 1、6、12 months after surgery.
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will evaluate the feasibility and effectiveness of urinary ctDNA detection and dynamic monitoring during treatment of NSCLC patients prospectively,by collecting and detecting tumor tissues, peripheral blood samples and urine samples of NSCLC patients.

DETAILED DESCRIPTION:
Liquid biopsy, specifically through the assessment of circulating tumor DNA(ctDNA) from peripheral blood, has shown great promise in lung cancer diagnosis and therapeutic monitoring.

Urinary samples are completely non-invasive and easily obtainable compared to blood and tissue extraction. To date, only a limited number of published studies have examined the feasibility of ctDNA detection from urine.

This study will collect tumor tissues, pretreatment peripheral blood samples and urine samples from different TNM stages of NSCLC patients, and detect EGFR gene mutations in paired samples.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 80 years
* Histologically confirmed diagnosis of stage non-small cell lung cancer undergoing surgical resection
* Completed and explicit information about TNM staging
* Paired specimens including tumor tissues, and both peripheral blood samples and urinary samples before and after surgery.
* Patients must have given written informed consent

Exclusion Criteria:

* Unable to comply with the study procedure
* Malignant tumor history within the past 5 years
* Coexisting small cell lung cancer
* Unqualified tissue, blood or urine samples

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Histologically confirmed stage non-small cell lung cancer patients with paired tumor tissue, peripheral blood samples, and urinary samples.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-06 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
The concordant frequency of genomic results among tumor tissue DNA, urinary ctDNA and peripheral blood ctDNA. | 12 months

SECONDARY OUTCOMES:
The difference of urine ctDNA detection effectiveness between different TNM stages NSCLC patients. | 18 months
Correlation of urine ctDNA concentration preoperative,intraoperative and 3 days after surgery with clinical features and prognosis. | 18 months
Lead time of tumor relapse detection by urine ctDNA than tumor markers and radiographic approaches. | 3 years
Urinary ctDNA predictive value for locoregional recurrence and distant metastasis. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Xiao Li, M.D, Study Director — Peking University People's Hospital
Locations (1):
- Peking University People'S Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
We will not make individual participant data (IPD) available

REFERENCES:
- [Background] Reckamp KL, Melnikova VO, Karlovich C, Sequist LV, Camidge DR, Wakelee H, Perol M, Oxnard GR, Kosco K, Croucher P, Samuelsz E, Vibat CR, Guerrero S, Geis J, Berz D, Mann E, Matheny S, Rolfe L, Raponi M, Erlander MG, Gadgeel S. A Highly Sensitive and Quantitative Test Platform for Detection of NSCLC EGFR Mutations in Urine and Plasma. J Thorac Oncol. 2016 Oct;11(10):1690-700. doi: 10.1016/j.jtho.2016.05.035. Epub 2016 Jul 25. PMID 27468937
- [Background] Su YH, Wang M, Brenner DE, Norton PA, Block TM. Detection of mutated K-ras DNA in urine, plasma, and serum of patients with colorectal carcinoma or adenomatous polyps. Ann N Y Acad Sci. 2008 Aug;1137:197-206. doi: 10.1196/annals.1448.027. PMID 18837947
- [Background] Lin SY, Dhillon V, Jain S, Chang TT, Hu CT, Lin YJ, Chen SH, Chang KC, Song W, Yu L, Block TM, Su YH. A locked nucleic acid clamp-mediated PCR assay for detection of a p53 codon 249 hotspot mutation in urine. J Mol Diagn. 2011 Sep;13(5):474-84. doi: 10.1016/j.jmoldx.2011.05.005. Epub 2011 Jul 2. PMID 21726666
- [Background] Janku F, Vibat CR, Kosco K, Holley VR, Cabrilo G, Meric-Bernstam F, Stepanek VM, Lin PP, Leppin L, Hassaine L, Poole JC, Kurzrock R, Erlander MG. BRAF V600E mutations in urine and plasma cell-free DNA from patients with Erdheim-Chester disease. Oncotarget. 2014 Jun 15;5(11):3607-10. doi: 10.18632/oncotarget.1964. PMID 25003820
- [Background] Hyman DM, Diamond EL, Vibat CR, Hassaine L, Poole JC, Patel M, Holley VR, Cabrilo G, Lu TT, Arcila ME, Chung YR, Rampal R, Lacouture ME, Rosen N, Meric-Bernstam F, Baselga J, Kurzrock R, Erlander MG, Janku F, Abdel-Wahab O. Prospective blinded study of BRAFV600E mutation detection in cell-free DNA of patients with systemic histiocytic disorders. Cancer Discov. 2015 Jan;5(1):64-71. doi: 10.1158/2159-8290.CD-14-0742. Epub 2014 Oct 16. PMID 25324352
- [Background] Crowley E, Di Nicolantonio F, Loupakis F, Bardelli A. Liquid biopsy: monitoring cancer-genetics in the blood. Nat Rev Clin Oncol. 2013 Aug;10(8):472-84. doi: 10.1038/nrclinonc.2013.110. Epub 2013 Jul 9. PMID 23836314